CLINICAL TRIAL: NCT03380494
Title: The Effectiveness of Overhead Perturbation Training on Joint Position Sense in Patients With Functional Shoulder Instability: A Pilot Study With Blinded, Randomized Controlled Trial Design
Brief Title: Overhead Perturbation Training for Glenohumeral Joint Instability
Acronym: OPT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 229780; 229780 (Registry Identifier: IRAS)
Record Dates: First submitted 2017-12-08; First posted 2017-12-21 (Actual); Last update posted 2018-02-20 (Actual); Status verified 2018-02

CONDITIONS: Exercise Movement Techniques; Shoulder Pain; Glenohumeral Subluxation
Keywords: Overhead perturbation training; instability, glenohumeral joint
MeSH Terms: conditions — Shoulder Pain; Shoulder Dislocation

STUDY DESIGN:
Intervention Model Description: Double blind, randomised controlled trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Overhead perturbation training technique (Experimental): Patients will undertake a series of exercise positions with the arm elevated above shoulder level with a stimulus applied with a weight and resistance band- such that the glenohumeral joint is exposed to a perturbed stimulus and has to utilise proprioception and motor control to correct arm position. The exercise session will be 45mins in length and occur once per week for 6 weeks.
  Interventions: Other: Overhead perturbation training
- Non-perturbed exercise (Active Comparator): Patients will undertake a series of exercise positions with the arm elevated above shoulder level with a stimulus applied via a weight held in the hand- such that the glenohumeral joint is exposed to a load but without a perturbation of joint position. The exercise session will be 45mins in length and occur once per week for 6 weeks.
  Interventions: Other: Non-perturbed training

INTERVENTIONS:
Other: Overhead perturbation training — A specifically chosen weight is attached to a 1m resistance band held above the head, hanging against gravity. The participant is encouraged to sustain a static position, where the weight and band provide variable magnitude perturbations to arm position. The body position of the participant is modified to facilitate greater and lesser perturbations. Bodily movements are prescribed to encourage joint perturbation. The participant undertakes 3 sets of 25 repetitions (60s rest) and continues with variable stimulus until fatigued.
  Other Names: OPT
  Arms: Overhead perturbation training technique
Other: Non-perturbed training — A weight is grasped by the participant and elevated above head to the same position as the OPT intervention. The participant is encouraged to sustain a static position. The body position of the participant is modified to facilitate greater and lesser perturbations. Bodily movements are prescribed to encourage joint perturbation. The participant undertakes 3 sets of 25 repetitions (60s rest) and continues with variable stimulus until fatigued.
  Arms: Non-perturbed exercise

SUMMARY:
The purpose of the trial is investigate the benefits of a novel, newly invented exercise technique protocol relative to physiological changes in upper limb proprioception (primary) and subjective readiness for return to sport (secondary).

The intervention (Overhead perturbation training) will be compared with a control intervention (non-perturbed stimulus) in a population of type II anterior glenohumeral joint instability patients (according to the Stanmore classification of instability). Each group will be assessed at baseline for glenohumeral joint proprioception (via lazer-pointer active relocation test), as well as perceived functional level (via Western Ontario Shoulder Instability index) and Shoulder Instability-Return to Sport after Injury (SIRSI) score. They will then undertake a 6 week exercise regime which is exactly the same- except the intervention used perturbated stimulus and the control uses non-perturbed stimulus. Outcome measures are re-assessed at the end of the intervention period. Results will be assessed statistically for statistical significance.

DETAILED DESCRIPTION:
Overhead athletic performance requires both static and dynamic mechanisms to coordinate glenohumeral and scapulothoracic stability to induce the appropriate motor response. Active function is predicated on a sufficient balance of muscular strength, endurance, flexibility and neuromuscular response to proprioceptive input. Coordinating, planning and synthesising complex multi-joint information is a process within the central nervous system, from the periphery to the higher centres of the brain, in a synergy of afferent and efferent feedback.

Joint position sense plays an important role for the shoulder joint in two key components of athletic performance: conscious limb placement and unconscious motor patterning in response to external force during movement. Such motor patterns can be characterised as the motor responsiveness to perturbations of joint position. This assists efficiency of muscular coordination when the shoulder is placed in the long lever position during overhead activities, where the desired motor pattern reaction is essential alongside contractile strength for successful performance and attenuation of injury risk. It is suggested that efficiency in neuromuscular control to provide responsive stabilization is necessary to sustain high levels of overhead performance and to avoid injury. The neuromuscular control response of the shoulder musculature on glenohumeral and scapulothoracic joint positions becomes deficient in the presence of structural injury. For example, rotator cuff injury specifically leads to deficiencies in neuromuscular control timing, patterning and strength compared with asymptomatic clients.

Perturbation of upper limb position during overhead activities causes unpredicted change in tissue length, resulting in a responsive pattern of muscular contractions. The OPT exercise series ensures that the deficient client is exposed to positions of vulnerability against displacement of the limb by external force. It is postulated that neural adaptations are induced through introduction of both rhythmic and sudden alterations to these positions A training stimulus (such as OPT) which facilitates neuromuscular control and speed of response to perturbation has potential to enhance overhead function. This signifies the role of neuromuscular control training in both rehabilitation and prevention of shoulder joint injury. The inclusion of this type of exercise training during rehabilitation and as part of injury risk minimisation strategies is an important component to sustain synchronization of muscular movement patterns.

Population in Focus

The subjects recruited for this study will be explained in greater depth further in the proposal, however are characterised by having a degree of functional glenohumeral joint instability. The physiotherapy class setting which will be utilised as the source of referrals is a heterogenous group of upper limb disorder patients, with a distinct sub group of individuals with functional instability who achieve sufficient recovery to meet the criteria for return to sport. According to the Stanmore classification of shoulder instability this group would correspond to Polar type II-III- that is placed on a continuum between atraumatic structural instability and non-structural, muscle patterning instability.

Current treatment versus OPT

The optimal management of anterior shoulder instability in those who undertake sport continues to be a challenge. Exercise therapy rehabilitation in a structured protocol shows statistically significant changes in validated outcome measures (Oxford Instability Shoulder Scores and Western Ontario Shoulder Index scores) but fails to incorporate exercise at the point of most instability through range of motion, particularly with sufficient challenge to the neuromuscular system to promote adaptation against perturbation at this point.

Of course OPT is not suggested to replace traditional measures of exercise therapy, but instead is designed to complement and optimise rehabilitation. By influencing both the physical and psychometric obstructions to return to activity, the OPT aims to improve patient care and enhance quality of life in its users. This has the additional benefit of streamlining the care pathway of this patient population, and in preparing them to return to higher levels of function, will potentially reduce recurrence of future injury. The pathway for these patients is optimised and made more efficient by providing the same amount of therapist contact, in a class setting to incorporate multiple users at once, but should enhance post intervention clinical scores. The application of similar programmes as a component of rehabilitation is already considered elsewhere; however the specific nature of OPT is suggested to enhance even these currently used protocols.

ELIGIBILITY:
Inclusion Criteria: A clinical presentation indicative of glenohumeral joint functional instability as classified by the Stanmore classification of shoulder instability Polar type II-III (on a continuum between atraumatic structural instability and non-structural, muscle patterning instability (Jaggi and Lambert, 2010)).

-

Exclusion Criteria:

* Presence of:
* Connective tissue disorder (Marfan's, Ehlos-Danlos)
* Nerve disorders: cervical radiculopathy +/- myotomal weakness; peripheral neuropathy/ palsy (long thoracic nerve palsy, axillary nerve palsy, suprascapular nerve palsy, etc.); brachial neuritis.
* Neuropathic peripheral sensitivity and/ or central sensitisation
* Post operative orthopaedic intervention < 12 weeks post MRI confirmed full thickness rotator cuff tear
* Distal upper limb/ hand pathology which limits the ability to grasp (including specific pathological signs of lateral epicondylaglia, carpal tunnel syndrome, carpal instability, etc).
* - inability to follow instructions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2018-04 (Estimated); Primary Completion 2018-06 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Lazer-pointer assisted angle relocation test | 6 weeks
  The laser pointer assisted angle-reproduction test (LP- ART) is a more simple and clinically friendly assessment tool. The outcome measure involves the patient pointing a wrist-mounted laser at 3 different targets (55', 90' and 125') in both the coronal and sagittal plane, with average of 3 being used. This method and has been shown to effectively quantify proprioceptive dysfunction in patients with shoulder instability (Balke, 2011).

SECONDARY OUTCOMES:
The Shoulder Instability-Return to Sport after Injury (SIRSI) score | 6 weeks
  The Shoulder Instability-Return to Sport after Injury (SIRSI) score has been developed and proposed as an easy to use score for evaluating an athlete's ability to return to sport. The score is validated and reliable in the use as an outcome measure for shoulder anterior instability patients (Gerometta et al. 2017).
Western Ontario Shoulder Instability Index (WOSI) | 6 weeks
  The tool is a patient completed, questionnaire consisting of 21 items, each scored on a 100mm Visual Analogue Scale (VAS). Each question is scored between 0-100 points and the summation of all the questions results in a final WOSI score. The final score ranges from 0 (best possible score - the patient is experiencing no decrease in shoulder-related quality of life) to 2100 (worst score - signifies extreme distress in shoulder-related quality of life).
  The WOSI is a valid, reliable and sensitive assessment for patients with shoulder problems that are associated with instability and it's widely recommended for use in the evaluation of these patients (Kirkley et al, 1998).

CONTACTS AND LOCATIONS:
Locations (1):
- Guys and St Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers.